CLINICAL TRIAL: NCT07269496
Title: An Open-label, Single-dose, Randomized, Two-way, Two-period Crossover Study to Compare Bioavailability and Pharmacokinetics of a Novel Furosemide Regimen Administered Subcutaneously Versus the Same Dose (80 mg) Administered Intravenously in Healthy Volunteers
Brief Title: Study to Compare Bioavailability and Pharmacokinetics of a Novel Furosemide Regimen Administered Subcutaneously Versus the Same Dose (80 mg) Administered Intravenously in Healthy Volunteers
Acronym: SQI-01-03
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SQ Innovation, Inc. (Industry)
Collaborators: BDD Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SQI-01-03; 1013098 (Other: IRAS)
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This study will be an open-label, single-dose, randomized, two-way, two-period crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SQIN-Furosemide is an investigational subcutaneous furosemide formulation at 30mg/mL (Experimental): In this study 80mg of SQIN-Furosemide will be administered subcutaneously over 5 hours using biphasic delivery profile of 30mg in the first hour and 50mg over the remaining 4 hours. IMP will be delivered by BD Alaris™ neXus CC Syringe Pump.
  Interventions: Drug: SQIN-Furosemide
- Sanofi Aventis 20mg/2mL Lasix infusion (Active Comparator): 80mg IV bolus administered over 2 doses of 40mg each for 10 mins, 2 hours apart (4mg/min).
  Interventions: Drug: Lasix ® Infusion

INTERVENTIONS:
Drug: SQIN-Furosemide — SQIN-Furosemide is a novel formulation of furosemide at 30mg/mL at pH 7.5 (range 7.1 to 7.8) intended for subcutaneous use.
  Other Names: Lasix ONYU
  Arms: SQIN-Furosemide is an investigational subcutaneous furosemide formulation at 30mg/mL
Drug: Lasix ® Infusion — Sanofi Aventis 20mg/2mL Lasix infusion. 80mg IV bolus administered over 2 doses of 40mg each for 10 mins, 2 hours apart (4mg/min).
  Other Names: Sanofi Aventis 20mg/2mL Lasix infusion
  Arms: Sanofi Aventis 20mg/2mL Lasix infusion

SUMMARY:
The trial is to compare the bioavailability of the original European Lasix (furosemide injection) administered in accordance with its prescribing information with the same dose of a novel furosemide formulation developed for this subcutaneous administration. The study will also investigate PK and PD of these regimens.

DETAILED DESCRIPTION:
This study will be an open-label, single-dose, randomized, two-way, two-period crossover study in 15 healthy adult volunteers.

Each participant will complete Screening, two Treatment phases, and Follow-up. The Screening Phase will be conducted on an outpatient basis up to 28 days prior to dosing. The Treatment Phase will comprise 2 crossover treatment periods separated by a minimum 7-day outpatient fluid re-equilibration and washout.

Participants will be admitted to the CRU on Day 1, and final eligibility assessments will be completed. Participants will be randomly assigned in a 1:1 ratio to 1 of 2 treatment sequences (AB or BA) to receive subcutaneous furosemide (Treatment A; Test) and IV furosemide (Treatment B; Reference). Participants randomized to sequence AB will receive subcutaneous furosemide for Treatment Period 1 and IV furosemide for Treatment Period 2, with treatments administered vice versa for sequence BA.

Study treatment based on the participant's assigned treatment sequence will be administered beginning in the morning of Day 1. SQIN-Furosemide will be administered by the BD Alaris™ neXus CC Syringe Pump and an infusion set programmed to delivers 30mg over first 60 minutes (total 1mL), followed by 50mg over 4 hours (total ~1.7mL), for a total dose and volume administered over 5 hours of 80mg and ~2.7mL, respectively. Furosemide Injection (20 mg/2mL) will be administered IV also with the use of the BD Alaris™ neXus CC Syringe Pump. Two doses of 40mg each will be infused at a rate of 4mg/min, such that the total amount of furosemide administered is 80 mg. PK, PD, and safety assessments will be collected over 24 hours, as detailed in the Schedule of Assessments. Participants will repeat the same procedures for Treatment Period 2 as for Treatment Period 1.

Participants will remain domiciled in the CRU through 24 hours after administration of study drug. Participants will be discharged from the CRU after all Day 2 study procedures and assessments have been completed, provided that safety parameters are acceptable to the Investigator. After the conclusion of Treatment 1 and prior to discharge, participants will be instructed regarding the diet and fluid intake, what to watch out for, how to contact study staff and when to return for Period 2. Participants will repeat the same procedures for Treatment Period 2 as for Treatment Period 1, this time receiving the alternative (cross-over) treatment.

Participants will be admitted to the CRU on the day of dosing in Treatment Period 2 and eligibility will be reconfirmed. subcutaneous or IV furosemide will then be administered on Day 9, according to the participant's randomization sequence, with PK, PD, and safety assessments collected over 24 hours, as detailed in the Schedule of Assessments.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female ≥18 years of age
* BMI between 18.5 and 32.0 kg/m2 (inclusive)
* Females will be non-pregnant and non-lactating
* Able to participate in the study in the opinion of the Investigator
* Has the ability to understand the requirements of the study and is willing to comply with all study procedures

Exclusion Criteria:

* Unable to consent to inclusion in study
* eGFR < 60 mL/min/1.73 m2
* Use of diuretics
* Systolic blood pressure (SBP) <90 mmHg
* Potassium < 3.5 or > 5.3 mmol/L
* Sodium < 133 or > 146 mmol/L
* Comorbidities or health issues which in the opinion of the investigator may interfere with study participation or study assessments.
* Major surgery within 30 days prior to Screening.
* Administration of an investigational drug or implantation of investigational device, or participation in another interventional trial, within 30 days prior to Screening, or 5 half-lives, whichever is longer.
* Pregnancy or breastfeeding
* Any contraindications for furosemide administration as per furosemide SmPC
* Any surgical or medical conditions, which in the opinion of the investigator may pose an undue risk to the participant, interfere with participation in the study or which may affect the integrity of the data
* Any clinically significant findings in Screening laboratory results which in the opinion of the investigator may pose an undue risk to the participant, interfere with participation in the study or which may affect the integrity of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Absolute bioavailability | From enrollment to end of treatment, 30 days
  Absolute bioavailability following 5-hour subcutaneous infusion based on a comparison of AUC (subcutaneous:IV) of furosemide.

SECONDARY OUTCOMES:
Pharmacokinetic parameters - Cmax | From beginning of treatment to 24 hours post-treatment
  Maximum plasma concentration (Cmax) over the timeframe of 24 hours
Urine volume | From beginning of treatment to 24 hours post-dose
  Urine volume in liters
Pharmacokinetic measures - Tmax | From beginning to 24 hours post-dose
  Time to Cmax (Tmax) over 24 hours
Pharmacokinetic measures - AUC | From beginning of treatment to 24 hours post-dose
  Area under the concentration versus time curve (AUC) from time 0 to the last measurable plasma concentration (AUClast) and to infinity (AUCinf), half-life (t½), apparent systemic clearance and volume of distribution (subcutaneous only), and systemic clearance and volume of distribution (IV only)
Sodium concentration in urine | From beginning of treatment to 24 hours post-dose
  Sodium concentration in urine in mmols

CONTACTS AND LOCATIONS:
Overall Officials: Lyn Cory, MD, Principal Investigator — BDD Pharma Ltd
Locations (1):
- BDD Pharma, Glasgow, Scotland, United Kingdom